CLINICAL TRIAL: NCT05236751
Title: Impact of Severe Intraoperative Hyperglycemia on Infection Rate After Elective Intracranial Interventions
Brief Title: Hyperglycemia in Neurosurgery
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: University of Roma La Sapienza (Other); Burdenko Neurosurgery Institute (Other)
Responsible Party: Sponsor
Other Study IDs: H-41050
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hyperglycemia; Postoperative Infection
Keywords: Intraoperative hyperglycemia; Postoperative infection; Neurosurgical patient; Open surgical intracranial intervention; Endoscopic intracranial intervention
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective intracranial intervention patients: Adult patients (18-89 years at the time of surgery) scheduled for elective intracranial (open surgical or endoscopic) intervention and require general anesthesia and a hospital stay of at least one day post-procedure.

SUMMARY:
Poor glycemic control is recognized as a risk factor for postoperative infection. For the neurosurgical patient, postoperative infection can lead to devastating complications such as meningitis, encephalitis and death. Neurosurgical patients often receive high doses of medications that increase blood glucose levels such as steroids, placing them at a potentially higher risk for postoperative infection. The purpose of this multisite observational study is to assess the impact of severe intraoperative hyperglycemia as a risk factor for postoperative infection in the neurosurgical patient.

DETAILED DESCRIPTION:
This is a multisite [3 locations] prospective observational study of adult patients (18-89 years old) scheduled for elective intracranial (open or endoscopic) procedures that require general anesthesia and a hospital stay of at least 1 day after the surgery. All sites will follow the standard of care clinical protocol for glycemic management that was developed at Boston Medical Center (BMC). Laboratory tests will be collected at the discretion of the primary clinician. This observational study does not require any change to routine clinical practice.

The following perioperative data (timeframe between Pre-Procedure Clinic visit through Post-Anesthesia Care Unit discharge): blood glucose measurements, total insulin dose, total dexamethasone dose, estimated intraoperative blood loss, antibiotic prophylaxis regimen.

The patient's electronic medical records data will be reviewed 7 days after the neurosurgical procedure to abstract all available culture data (blood, urine, sputum, CSF), available treatment regimen data prescribed for infection (antibiotics), complications from hyperglycemia (diabetic ketoacidosis, hyperglycemic nonketotic coma) or insulin therapy (hypoglycemia episodes). Intensive care unit (ICU) and hospital length of stay will also be obtained form the medical records.

The investigators anticipate finding four groups of patients with regards to intraoperative blood glucose levels and management: 1) patients with no episodes of severe intraoperative hyperglycemia, 2) patients with intraoperative hyperglycemia who received insulin treatment, 3) patients with intraoperative hyperglycemia who did not receive insulin treatment and 4) patients with no available laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective intracranial (open surgical or endoscopic) intervention
* General anesthesia
* Hospital stay of at least 1 day post-procedure

Exclusion Criteria:

* Diagnosis of infection (local or systemic) in preoperative period
* Emergency procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-89 years at the time of surgery) scheduled for elective intracranial (open surgical or endoscopic) intervention and require general anesthesia and a hospital stay of at least 1 day post-procedure.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Postoperative infection | 7 days after surgery
  Proportion of patients diagnosed with infection (such as wound, pulmonary, urological, blood) in the postoperative period

SECONDARY OUTCOMES:
Antibiotic prophylaxis scheme | Preoperatively
  Types of antibiotics administered preoperatively abstracted from electronic medical records.
Intraoperative glucose level in whole blood | before incision and at the end of surgery
  Twice intraoperatively abstracted from electronic medical records
Intraoperative dose of insulin | During surgical procedure
  Abstracted from electronic medical records
Dosages and regimen of dexamethasone in the perioperative period | preoperative clinic visit to within 7 days of surgery
  Abstracted from electronic medical records
Perioperative complications | preoperative clinic visit to within 7 days of surgery
  Perioperative complications (such as episodes of hemodynamic instability, blood loss) abstracted from electronic medical records
Duration of stay in ICU in hours | 30 days
  Abstracted from electronic medical records
Duration of stay in hospital in days | 30 days
  Abstracted from electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Canelli, MD, Principal Investigator — Boston Medical Center
Locations (3):
- Boston Medical Center, Boston, Massachusetts, United States
- Sapienza University, Rome, Italy
- Burdenko Neurosurgery Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided